CLINICAL TRIAL: NCT00991718
Title: A Phase I, Open-Label Absorption, Distribution, Metabolism, and Excretion (ADME) Study of the Hedgehog Pathway Inhibitor GDC-0449 in Healthy Female Subjects of Non-Childbearing Potential
Brief Title: A Study of the Hedgehog Pathway Inhibitor GDC-0449 in Healthy Female Subjects of Non-Childbearing Potential
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SHH4683g
Record Dates: First submitted 2009-10-06; First posted 2009-10-08 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Healthy
Keywords: GDC0449
MeSH Terms: interventions — HhAntag691; Product Labeling

ARMS (4):
- A (Experimental): On Day 1, subjects received a single oral dose of non-labeled GDC-0449 and a single IV tracer dose of 14C-GDC-0449.
  Interventions: Drug: GDC-0449 oral capsules (non-labeled); Drug: GDC-0449 IV injection (labeled)
- B (Experimental): On Day 1, subjects received a single oral dose of 14C-GDC-0449.
  Interventions: Drug: CDC-0449 oral suspension (labeled)
- C (Experimental): On Days 1-7, subjects received a single oral dose of non-labeled GDC-0449. On Day 7, subjects also received a single IV tracer dose of 14C-GDC-0449.
  Interventions: Drug: GDC-0449 oral capsules (non-labeled); Drug: GDC-0449 IV injection (labeled)
- D (Experimental): On Days 1-6, subjects received a single oral dose of non-labeled GDC-0449. On Day 7, subjects received a single oral dose of 14C-GDC-0449.
  Interventions: Drug: GDC-0449 oral capsules (non-labeled); Drug: CDC-0449 oral suspension (labeled)

INTERVENTIONS:
Drug: GDC-0449 oral capsules (non-labeled) — 150 mg oral capsule
  Arms: A; C; D
Drug: GDC-0449 IV injection (labeled) — 10 mcg (in 2 mL) IV dose of 14C-GDC-0449
  Arms: A; C
Drug: CDC-0449 oral suspension (labeled) — 30-mL oral suspension containing 6.5 mcg 14CGDC-0449 and 150 mg GDC-0449
  Arms: B; D

SUMMARY:
This is an open-label, Phase I, single-center, single-dose administration study to determine the absolute bioavailability, clearance, and volume of distribution of GDC-0449 (Part A) and to determine the routes of excretion and extent of metabolism of GDC-0449 (Part B). Parts A and B will be conducted sequentially, with ≥ 7 days between dosing the sixth subject in Part A and dosing the first subject in Part B. In each part, 6 healthy female subjects of non-childbearing potential, between 18 and 65 years of age (inclusive), will be dosed.

ELIGIBILITY:
Inclusion Criteria

* Female
* Non-childbearing potential
* Body mass index (BMI) between 18 and 32 kg/m^2, inclusive
* In good health, determined by no clinically significant findings on physical examination, medical history, 12-lead ECG, and vital signs
* Negative test for drugs of abuse at screening (does not include alcohol) and at admission to the clinical research facility (does include alcohol)

Exclusion Criteria

* History or clinical manifestations of clinically significant metabolic, hepatic, renal, hematologic, pulmonary, cardiovascular, endocrine, gastrointestinal (including gastric or duodenal ulcers), urologic, neurologic, inflammatory, or psychiatric disorders, or cancer
* History of symptomatic hypotension, idiopathic orthostatic hypotension, or other autonomous-failure syndromes
* History of severe physical injury, direct impact trauma, or neurological trauma within 6 months prior to Day -1
* History of stomach or intestinal surgery, stomach disease, or resection that would potentially alter absorption and/or excretion of orally administered drugs (appendectomy, hernia repair, and/or cholecystectomy are allowed)
* History of alcoholism, drug abuse, or drug addiction (including soft drugs like cannabis products)
* Use of any prescription medications/products, including known enzyme-inducing/inhibiting agents, over-the-counter medication, or other non-prescription preparations (including supplements, vitamins, minerals, phytotherapeutic/herbal/ plant-derived preparations, the tryptophans, and St. John's wort or other hypericum perforatum-containing substance) within 2 weeks prior to Day -1, with the exception of hormone-replacement therapy
* Participation in any other investigational drug study in which receipt of an investigational study drug occurred within 60 days prior to Day -1 or within 5 times the elimination half-life of the respective drug; participation in a trial involving administration of ^1^4C-radiolabeled compound(s) within 6 months prior to Day -1; participation in more than two other drug trials within 1 year prior to Day -1
* Receipt of any vaccination or immunization within 1 month prior to Day -1
* Use of any nicotine-containing or nicotine-replacement products within 6 months prior to Day -1
* Consumption of alcohol or methylxanthine-containing beverages or food
* Receipt of blood products within 2 months prior to Day -1
* Donation of > 100 mL of blood within 60 days prior to Day -1; donation of > 1.0 litres of blood within 10 months prior to Day -1
* Irregular defecation pattern, i.e., less than once per 2 days within 6 months prior to Day -1; acute constipation problems within 3 weeks prior to Day -1 (Part B subjects only)
* Poor peripheral venous access

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
PK (Max observed and time to max plasma concentrations, area under the plasma concentration-time curve, absolute bioavailability, total plasma clearance, vol of dist, plasma terminal phase half-life, cumulative % excretion in urine and feces [Part B]) | Until study discontinuation

SECONDARY OUTCOMES:
Safety outcome measures (incidence, nature, and severity of adverse events; change in clinical laboratory results; change in vital signs; change in electrocardiogram [ECG]; and change in physical examination findings) | Until study discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Low, M.D., Study Director — Genentech, Inc.